CLINICAL TRIAL: NCT04497259
Title: Using Tele-evaluation and Teleconsultation Instead of Classical Consultation for the Follow-up of Obese Patients After Bariatric Surgery : a Pilot Study.
Brief Title: Follow-up of Bariatric Surgery by Teleconsultations
Acronym: TELECHIRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/19/0128
Record Dates: First submitted 2020-02-10; First posted 2020-08-04 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: bariatric surgery; follow-up; tele-evaluations; e-medicine
MeSH Terms: conditions — Obesity | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): Patients in the teleconsultation arm will benefit from a tele-evaluation (a questionnaire filled through a chatbot link) and teleconsultation (skype-like connection) at 6 and 9 months after surgery.
  Interventions: Other: Teleevaluation; Other: Teleconsultation
- Control (Experimental): Patients in the consultation arm will benefit from a tele-evaluation (a questionnaire filled at home after the file was sent by secured mail) and a classical face to face consultation at 6 and 9 months after surgery.
  Interventions: Other: Teleevaluation; Other: Classical consultation

INTERVENTIONS:
Other: Teleevaluation — Patients will answer to a questionnaire filled through a chatbot link
Other: Teleconsultation — A teleconsultation (skype-like connection) at 6 and 9 months after surgery
  Arms: Interventional
Other: Classical consultation — Patients in the consultation arm will benefit from a classical face to face consultation at 6 and 9 months after surgery.
  Arms: Control

SUMMARY:
An organised follow-up is required after bariatric surgery, but 50% of patients are lost to follow-up after 2 years. To design a large randomized clinical trial (RCT) comparing teleevaluations and teleconsultations to classical follow, aiming to prove that the quality of the follow-up is maintained and the patient-experience is improved, at a lower cost in people living far from the reference centre, this pilot study aims at describing the distribution of the collected criteria.

DETAILED DESCRIPTION:
An organised follow-up is required after bariatric surgery, but 50% of patients are lost to follow-up after 2 years. This follow-up requires about 5 multi-professional evaluations during the first year. This can be cumbersome in patients living far from the reference centre and who may perceive the necessary time, cost and lost of income, and constraints as imbalanced. Teleevaluations and teleconsultations may solve this issue by replacing some of the classical evaluations (at 6 and 9 months). An RCT would be necessary, and a pilot study is proposed to describe the distribution of the judgment criteria.

This pilot study aims at describing all the parameters necessary to build an RCT, and involves the randomisation of operated patients recruited 3 months after surgery, in to groups. One will have the classical follow-up (venue and consultations at 6 and 9 months) the over will have teleevaluations and teleconsultations ; the parameters will be described at 12 months. The teleevaluation is either proposed as usual (a file is sent by secure mail) or by chatbot interaction. The consultation and the teleconsultation are based on the standard of care scenario.

ELIGIBILITY:
Inclusion Criteria:

* adults having had bariatric surgery 3 months before
* able to use an internet tool of chatbot and skype-like secured connection
* adult under 60 years old
* free inform and sign consent
* living more than 50km from Toulouse
* persons with social security

Exclusion Criteria:

* complications at the 3rd month post-surgery requiring specific care
* insufficient internet connection
* minor
* pregnant women
* protected adults
* people in emergency
* people unable to give consent

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-02-26 (Estimated); Study Completion 2025-02-26 (Estimated)

PRIMARY OUTCOMES:
Composite score research | month 12
  Look for the composite follow-up quality score taking into account weighting results, co-morbidities, absence of complications and skill acquisition.

SECONDARY OUTCOMES:
Coefficient evaluation | month 12
  Coefficient of variation and Cronbach's coefficient assessing the quality of the composite follow-up quality score
Consultation measure | month 6 and 9
  the time of a teleconsultation and a face-to-face consultation, by an objective measurement of this time at 6 and 9 months postoperatively
Composite distribution | month 12
  the distribution of each of the components of the Composite Follow-up Quality Score in the two arms of the study
Consultation feeling | Month 6 and 9
  satisfaction and constraints felt with regard to teleconsultations, by scores measured at teleconsultations and consultation at 6 and 9 months post-operatively
Consultation feasability | month 6 and 9
  the feasibility of teleconsultation and consultation with scores measured at 6 and 9 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Patrick RITZ, Md, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Ritz, Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No